CLINICAL TRIAL: NCT05044650
Title: A Study to Evaluate the Efficacy of KOVIR Capsule (TD0069) in the Combination Regimen With Background Treatment in COVID-19 Patients Without Symptoms of Acute Respiratory Distress
Brief Title: Efficacy of KOVIR Capsule in the Combination Regimen With Background Treatment in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YDHDT-KOVIR-B
Record Dates: First submitted 2021-09-13; First posted 2021-09-16 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be assigned randomly 7:3 to either KOVIR group or Non-KOVIR group respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KOVIR (Experimental): Standard dose, 3 capsules/time x 3 times/day x 14 days combined with background treatment
  Interventions: Dietary Supplement: KOVIR capsule combined with background treatment
- NON-KOVIR (No Intervention): Only background treatment

INTERVENTIONS:
Dietary Supplement: KOVIR capsule combined with background treatment — KOVIR is a hard capsule containing fine powder mixed medicinal herbs 600 mg
  Arms: KOVIR

SUMMARY:
The acute pneumonia pandemic caused by a new strain of corona virus 2019, namely as COVID-19 by the World Health Organization (WHO), is a pandemic caused by SARS-CoV-2 virus. The reported symptoms vary from fever or chills, cough, shortness of breath, to muscle aches, headaches, loss of taste or smell.

The capsule KOVIR is a product based on the traditional medicine named "Ren shen bai du san" which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

DETAILED DESCRIPTION:
The acute pneumonia pandemic caused by a new strain of corona virus 2019, namely as COVID-19 by the World Health Organization (WHO), is a pandemic caused by SARS-CoV-2 virus. The reported symptoms have included, but are not limited to fever or chills, cough, shortness of breath, muscle aches, headaches, loss of taste or smell, diarrhea, dizziness, sore throat, abdominal pain, anorexia, and vomiting.

The capsule KOVIR is a product based on the traditional prescription named "Ren shen bai du san" which is used to treat the cold conditions, also known as the initial plague according to the theory of traditional medicine.

The study compares between standard dose regimen of KOVIR combined with background treatment in COVID-19 patients and only background treatment in COVID-19 patients. The study will enroll 700 participants to KOVIR group and 300 participant to Non-KOVIR group.

All participants will be treated and followed up in 14-day period. In case the participant meets the discharge criteria before 14 days, discontinuing the study drug will be done at the discretion of the investigators.

Screening procedures occur at Day 1. Periodic assessments are conducted daily from Day 2-14. Finally, End of study visit is conducted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18-65, Vietnamese nationality
* Participants diagnosed with Positive result of SARS-CoV-2 using real time RT-PCR test, Ct value <30 (equivalent to viral load > 3log)
* Voluntary participation in the study by signing an informed consent
* Ability to adhere to treatment according to the investigator's assessment

Exclusion Criteria:

* Symptoms of severe upper and lower respiratory tract infections such as dyspnea, SpO2<93%.
* Acute reduction of ventilation function of respiratory apparatus and/or respiration function of the lung in any of the following three groups:

  * Respiratory distress due to hypoxemia with PaO2 less than 60mmHg when breathing room air.
  * Respiratory distress due to hypercapnia with PaCO2 above 50mmHg
  * Mixed respiratory distress accompanied by both a decrease in PaO2 and an increase in PaCO2
* Allergy/intolerance to any component of the study drug.
* Inability to administer medicine.
* Severe pneumonia as assessed by the investigator.
* Inability to comply with study procedures or to ensure compliance with study drug administration as assessed by investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Mean duration of clinical symptoms | up to 14 days
  Mean time from baseline to no clinical symptom of COVID-19
Number of participants with respiratory distress complications requiring treatment | up to 14 days
  Occurrence of symptoms of respiratory distress complications requiring treatment
Change in the severity of daily symptoms | up to 14 days
  Scale: 0 = Asymptomatic, 1 = Mild, 2 = Moderate, 3 = Severe
Number of Participants with Adverse Events as Assessed by CTCAE v5.0 | up to 30 days after last dose
  Frequency and severity of Study drug-related adverse events, adverse events leading to study termination, serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Loc Huynh, SL II., MD., Principal Investigator — Traditional Medicine Institute in Ho Chi Minh City
Locations (1):
- Traditional Medicine Institute in Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No